CLINICAL TRIAL: NCT00454129
Title: ERC Via Double-Balloon-Enteroscopy in Patients With Biliodigestive Anastomosis
Acronym: DBE ERC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Heidelberg University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: DBE ERC
Record Dates: First submitted 2007-03-29; First posted 2007-03-30 (Estimated); Last update posted 2013-01-28 (Estimated); Status verified 2007-03

CONDITIONS: Cholangiography
Keywords: Feasibilty of cholangiography via double-balloon enteroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: cholangiography via double-balloon enteroscopy
Procedure: MR cholangiography

SUMMARY:
In patients with biliodigestive anastomosis direct cholangiography (ERC) is due to changed anatomy commonly not possible. The aim of the study is to test the feasibility to perform direct cholangiography in these patients via double-balloon enteroscopy and to compare it to MR cholangiography.

ELIGIBILITY:
Inclusion Criteria:

* Biliodigestive anastomosis; and
* Suspicion of biliary disorder

Exclusion Criteria:

* Exclusion criteria of double-balloon enteroscopy and MR-cholangiography

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2007-03

CONTACTS AND LOCATIONS:
Overall Officials: Jens Encke, Prof., Principal Investigator — Medical University of Heidelberg
Locations (1):
- Medical University of Heidelberg, Department of Gastroenterology, Heidelberg, Germany